CLINICAL TRIAL: NCT04327726
Title: Effectiveness of Nebulized Dexmedetomidine for Treatment of Post-Dural Puncture Headache in Parturients Undergoing Elective Cesarean Section Under Spinal Anesthesia: Randomized Controlled Study
Brief Title: Effectiveness of Nebulized Dexmedetomidine for Treatment of Obstetric Post-Dural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6075-26-4-2020
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be aware of their group assignment, and the medications will be prepared by an anesthetist who is not involved in the study. The anesthetist who will assess the participants after the intervention is blinded to the group allocation and single experienced operator who is unaware of patient group and study purpose will perform all Trans-Cranial Doppler (TCD) measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): received ultrasonic nebulization of 4mL 0.9% saline twice daily for 3 days
  Interventions: Other: 0.9% Saline Nebulization
- Dexmedetomidine group (Active Comparator): received ultrasonic nebulization of 1 µg/kg dexmedetomidine diluted in 4mL 0.9% saline twice daily for 3 days. The intervention will be continued until achieving a VAS score ≤3 and Lybecker et al. classification score <2 and or for a maximum of 72 hours. Patients in this group who achieved the target scores before 72 hours will be given 4ml of saline 0.9% nebulization to maintain blinding.
  Interventions: Drug: Dexmedetomidine Nebulization

INTERVENTIONS:
Drug: Dexmedetomidine Nebulization — ultrasonic nebulization of 1 µg/kg dexmedetomidine for PDPH treatment
  Arms: Dexmedetomidine group
Other: 0.9% Saline Nebulization — nebulization of 4mL 0.9% saline
  Arms: Control group

SUMMARY:
Postdural puncture headache (PDPH) is a common complication, following neuraxial techniques. The obstetric population is particularly prone to PDPH. Therefore, treatment of PDPH is a key issue in obstetric anesthesia.

Dexmedetomidine is a highly selective, centrally acting α2-adrenergic agonist with analgesic and anxiolytic effects. Moreover, it decreases cerebral blood flow (CBF) in humans and animals secondary to cerebrovascular vasoconstriction. It has been used via the intranasal and inhalational routes for many purposes including premedication, sedation and postoperative analgesia. Because of its desirable properties, we hypothesized that dexmedetomidine nebulization could be effective in the treatment of patients suffering from PDPH after caesarean section.

DETAILED DESCRIPTION:
Post-Dural puncture headache (PDPH) is a well-known common devastating complication of subarachnoid block. Despite the decreasing incidences of PDPH over the last years due to the advancement in the design and smaller size of spinal needles, PDPH remains to be a common complication in post-partum patients. Female gender, typically pregnant females, young age, low body mass index, dilutional anemia, and the preference of neuraxial anesthesia for Cesarean Section renders obstetric patients to be more exposed to PDPH. Consequently, treating this complication is of paramount importance in obstetric anesthesia.

The cause of PDPH is not entirely known but there is a considerable evidence support the explanation of the low cerebrospinal fluid (CSF) pressure resulting from continuous CSF leak through the tear in meninges that exceeds the CSF production rate as a main cause of PDPH. As little as 10% CSF volume loss could induce PDPH from the traction on the pain sensitive intracranial structures in the upright position combined with reflex vasodilatation. Several treatment options have been proposed which are usually consisting of bed rest in supine position, fluid therapy, analgesics, sumatriptan and caffeine. Epidural blood patch remained the gold standard therapy but it is an invasive technique.

Dexmedetomidine (Dex) is a highly selective centrally acting α2-adrenoreceptor agonist that produces cooperative sedation, anxiolysis, and analgesia with minimal respiratory depression. Moreover it was found to attenuate the stress and inflammatory response to anesthetic and surgical procedures. Stimulation of α2-receptors in substantia gelatinosa of the dorsal horn leads to suppression of nociceptive neurons firing and inhibition of substance-P release also, its stimulation in the locus coeruleus area which is known to be a significant nociceptive transmission modulator terminates pain signals transmission resulting in analgesia. Additionally, an existing literature supports that Dex decreases cerebral blood flow (CBF) in humans and animals secondary to cerebrovascular vasoconstriction. Thus, the use of Dex might be a useful adjunct in certain situations that require cerebral vasoconstriction together with analgesia such as PDPH. The present study will be undertaken to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Post-partum females diagnosed with PDPH after elective caesarean section under spinal anesthesia and with visual analogue score (VAS) ≥ 4 and Lybecker et al. classification score ≥2.
* Age 21- 40 years old.
* ASA I and ASA II.
* Accepted mental state of the patient.

Exclusion Criteria:

* Patient refusal.
* ASA Grade III and IV.
* Emergent caesarean section.
* Inadequate temporal window.
* Hypertensive disorders of the pregnancy.
* Atrial fibrillation.
* History of allergy to local anesthetics.
* History of chronic headache, migraine, convulsions, and cerebrovascular accident.
* Contraindication to spinal anesthesia: coagulopathy, infection at site of injection

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
visual analogue score (VAS) | 24 hour
  using the 10-cm visual analogue score (VAS) where score 0 is no headache and 10 is the worst imaginable headache with 1-3 classified as mild, 4-6 moderate, and 7-10 severe our aim to get VAS </= 3 at 24 hour from starting treatment
Lybecker headache classification score | 24 hour
  our aim to get Lybecker score < 2 at 24hour following treatment Lybecker et al. classification of PDPH score 1: Mild PDPH where daily activities slightly restricted. Patient is not bedridden.
  No associated symptoms*. Score 2:Moderate: Daily activities significantly restricted and most of the day patient is bedridden with or without associated symptoms.
  Score 3:Severe Daily activities completely restricted, patient is bedridden all the day and always with associated symptoms Associated symptoms include: Nausea, vomiting, vertigo, dizziness, tinnitus Photophobia, diplopia, and neck stiffness.

SECONDARY OUTCOMES:
the effects of nebulized dexmedetomidine on cerebral blood flow by using Trans-Cranial Doppler (TCD) | 72 hours
  TCD measurements (mean flow velocity, pulsatility index) will be performed at 0, 24, 48, 72hours
adverse effects related to nebulized Dexmedetomidine | 72 hours
  occurrence of any adverse effects (Hypotension, bradycardia, sedation) related to nebulized Dexmedetomidine

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University; Shereen E Abd Ellatif, MD, Study Director — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the individual participant data and any additional supporting information will become available starting 6 months after publication.
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Sachs A, Smiley R. Post-dural puncture headache: the worst common complication in obstetric anesthesia. Semin Perinatol. 2014 Oct;38(6):386-94. doi: 10.1053/j.semperi.2014.07.007. Epub 2014 Aug 19. PMID 25146108
- [Background] Bardon J, LE Ray C, Samama CM, Bonnet MP. Risk factors of post-dural puncture headache receiving a blood patch in obstetric patients. Minerva Anestesiol. 2016 Jun;82(6):641-8. Epub 2015 Jul 29. PMID 26222393
- [Background] FitzGerald S, Salman M. Postdural puncture headache in obstetric patients. Br J Gen Pract. 2019 Apr;69(681):207-208. doi: 10.3399/bjgp19X702125. No abstract available. PMID 30923161
- [Background] Shah A, Bhatia PK, Tulsiani KL. Post dural puncture headache in caesarean section-a comparative study using 25G Quincke, 27G Quincke and 27G Whitacre needle. Indian J Anaesth 2002; 46(5):373-377.
- [Background] Turnbull DK, Shepherd DB. Post-dural puncture headache: pathogenesis, prevention and treatment. Br J Anaesth. 2003 Nov;91(5):718-29. doi: 10.1093/bja/aeg231. PMID 14570796
- [Background] Amorim JA, Gomes de Barros MV, Valenca MM. Post-dural (post-lumbar) puncture headache: risk factors and clinical features. Cephalalgia. 2012 Sep;32(12):916-23. doi: 10.1177/0333102412453951. Epub 2012 Jul 27. PMID 22843225
- [Background] Uyar Turkyilmaz E, Eryilmaz NC, Guzey NA, Moraloglu O. [Bilateral greater occipital nerve block for treatment of post-dural puncture headache after caesarean operations]. Rev Bras Anestesiol. 2016 Sep-Oct;66(5):445-50. doi: 10.1016/j.bjan.2015.12.001. Epub 2016 Jul 18. Portuguese. PMID 27445257
- [Background] Tsaousi GG, Bilotta F. Is dexmedetomidine a favorable agent for cerebral hemodynamics? Indian J Crit Care Med. 2016 Jan;20(1):1-2. doi: 10.4103/0972-5229.173675. No abstract available. PMID 26955209
- [Background] Tang C, Huang X, Kang F, Chai X, Wang S, Yin G, Wang H, Li J. Intranasal Dexmedetomidine on Stress Hormones, Inflammatory Markers, and Postoperative Analgesia after Functional Endoscopic Sinus Surgery. Mediators Inflamm. 2015;2015:939431. doi: 10.1155/2015/939431. Epub 2015 Jun 25. PMID 26199465
- [Background] Jaakola ML, Salonen M, Lehtinen R, Scheinin H. The analgesic action of dexmedetomidine--a novel alpha 2-adrenoceptor agonist--in healthy volunteers. Pain. 1991 Sep;46(3):281-285. doi: 10.1016/0304-3959(91)90111-A. PMID 1684653
- [Background] Gertler R, Brown HC, Mitchell DH, Silvius EN. Dexmedetomidine: a novel sedative-analgesic agent. Proc (Bayl Univ Med Cent). 2001 Jan;14(1):13-21. doi: 10.1080/08998280.2001.11927725. PMID 16369581
- [Background] Gerlach AT, Dasta JF. Dexmedetomidine: an updated review. Ann Pharmacother. 2007 Feb;41(2):245-52. doi: 10.1345/aph.1H314. Epub 2007 Feb 13. Erratum In: Ann Pharmacother. 2007 Mar;41(3):530-1. PMID 17299013
- [Background] Drummond JC, Dao AV, Roth DM, Cheng CR, Atwater BI, Minokadeh A, Pasco LC, Patel PM. Effect of dexmedetomidine on cerebral blood flow velocity, cerebral metabolic rate, and carbon dioxide response in normal humans. Anesthesiology. 2008 Feb;108(2):225-32. doi: 10.1097/01.anes.0000299576.00302.4c. PMID 18212567
- [Background] Kumar A, Kumar A, Sinha C, Anant M, Singh JK. Dexmedetomidine nebulization: an answer to post-dural puncture headache? Int J Obstet Anesth. 2019 Nov;40:155-156. doi: 10.1016/j.ijoa.2019.06.004. Epub 2019 Jun 19. No abstract available. PMID 31345663
- [Background] Lybecker H, Djernes M, Schmidt JF. Postdural puncture headache (PDPH): onset, duration, severity, and associated symptoms. An analysis of 75 consecutive patients with PDPH. Acta Anaesthesiol Scand. 1995 Jul;39(5):605-12. doi: 10.1111/j.1399-6576.1995.tb04135.x. PMID 7572008
- [Background] Bathala L, Mehndiratta MM, Sharma VK. Transcranial doppler: Technique and common findings (Part 1). Ann Indian Acad Neurol. 2013 Apr;16(2):174-9. doi: 10.4103/0972-2327.112460. PMID 23956559
- [Derived] Mowafy SMS, Ellatif SEA. Effectiveness of nebulized dexmedetomidine for treatment of post-dural puncture headache in parturients undergoing elective cesarean section under spinal anesthesia: a randomized controlled study. J Anesth. 2021 Aug;35(4):515-524. doi: 10.1007/s00540-021-02944-6. Epub 2021 May 16. PMID 33993346